CLINICAL TRIAL: NCT04527510
Title: Remote Breast Cancer Screening Based on Automated Breast Ultrasound Among Chinese Women: a Multi-center, Prospective, Cohort Study
Brief Title: Remote Breast Cancer Screening Study
Status: Active, not recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of the Fourth Military Medical University (Other)
Responsible Party: Principal Investigator, Song Hongping, Principal Investigator, The First Affiliated Hospital of the Fourth Military Medical University
Other Study IDs: 2021LC2210
Record Dates: First submitted 2020-08-23; First posted 2020-08-26 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Mass Screening; Cancer Screening; Ultrasound Imaging; AI (Artificial Intelligence)
Keywords: Remote breast cancer screening; AB US; AI; Scanning and reading patterns
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Conventional-reading
  Interventions: Diagnostic Test: Conventional-reading
- Second-reading
  Interventions: Diagnostic Test: Second-reading
- Concurrent-reading
  Interventions: Diagnostic Test: Concurrent-reading
- Tow-view-reading
  Interventions: Diagnostic Test: Tow views-reading
- Handheld US-screening
  Interventions: Diagnostic Test: Handheld US-screening

INTERVENTIONS:
Diagnostic Test: Conventional-reading — Two radiologists interpret at least three views of each breast without AI independently.
  Groups: Conventional-reading
Diagnostic Test: Second-reading — One radiologist reads AB US images without AI first, then combines the indications of AI marks to make the final decision.
  Groups: Second-reading
Diagnostic Test: Concurrent-reading — One radiologist identifies CAD marks first, then quickly browses the entire AB US examination to make the final decision.
  Groups: Concurrent-reading
Diagnostic Test: Tow views-reading — Two radiologists interpret only two views of each breast without AI independently.
  Groups: Tow-view-reading
Diagnostic Test: Handheld US-screening — One radiologist screens the breast cancer using Handheld US and interprets images immediately.
  Groups: Handheld US-screening

SUMMARY:
A multi-center, prospective, cohort study to evaluate the efficiency of breast cancer screening based on Automated Breast Ultrasound (AB US) with remote reading mode.

DETAILED DESCRIPTION:
The burden of breast cancer incidence and mortality is rapidly growing during the past two decades in China. Screening has been proven to be effective in detecting early-stage disease and reducing mortality of 10% to 39% due to breast cancer. US is used as a primary screening method among Chinese women because Asian women characteristically have higher-density breasts than other ethnic groups. However, US is dependent on operator experience, lack of standardized scanning protocols, limited ultrasound physician and heavy workloads. In order to improve the efficiency and quality of breast cancer screening among Chinese women, a new remote screening pattern based on AB US was proposed and studied for breast cancer in China. This multi-center, prospective, cohort study aims to evaluate the efficiency of breast cancer screening based on AB US with remote reading mode. In addition, we will also explore the practice value of AI on AB US screening and efficient image acquiring and reading modes of AB US.

ELIGIBILITY:
Inclusion Criteria:

1. Any age at 35 and over
2. Screening breast cancer with AB US
3. Obtaining written informed consent

Exclusion Criteria:

1. symptoms of breast cancer
2. surgical of breast within 12 months prior to the study
3. known diagnosis breast cancer
4. poor image quality
5. follow-up was less than 12 months

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 5714 women are needed (at least 12 cancer cases are expected with 80% power and 20% dropout)
Sampling Method: Probability Sample
Enrollment: 6333 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The performance of breast cancer screening based on AB US with remote reading mode | 4 years
  The performance of breast cancer screening based on AB US with remote reading mode will be evaluated by cancer detection rate, recall rate, sensitivity, specificity, positive predictive value, early detection of breast cancer, interval cancers and time for image acquisition and interpretation.

SECONDARY OUTCOMES:
Evaluate the performance of AI on breast cancer screening based on AB US with remote reading mode | 4 years
  Evaluate the performance of AI on breast cancer screening based on AB US with remote reading mode (Conventional-reading vs. Second-reading / Concurrent-reading)
Evaluate the performance of the image acquisition and interpretation modes in breast cancer screening based on AB US with remote reading mode | 4 years
  Evaluate the performance of the image acquisition and interpretation modes in breast cancer screening based on AB US with remote reading mode (two views vs. three views)
Evaluate the performance of breast cancer screening according to the breast US device | 4 years
  Evaluate the performance of breast cancer screening according to the breast US device (Hand-held US vs. AB US)

CONTACTS AND LOCATIONS:
Overall Officials: Hongping Song, PHD,MD, Principal Investigator — Xijing hospital of The fourth military medical university
Locations (2):
- China (2):
  - The First Affiliated Hospital of Fourth Military Medical University, Xi'an, Shaanxi
  - The First Affiliated Hospital of the Fourth Military Medical University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dang X, Gao Y, Ju Y, Yuan X, Lin H, Ren Y, Xiao Y, Shu R, Gu X, Moon WK, Song H. Automated Breast Ultrasound With Remote Reading for Primary Breast Cancer Screening: A Prospective Study Involving 46 Community Health Centers in China. AJR Am J Roentgenol. 2025 Jan;224(1):e2431830. doi: 10.2214/AJR.24.31830. Epub 2024 Oct 23. PMID 39440797